CLINICAL TRIAL: NCT04284800
Title: Evaluation of Potential Myocardial Injury in Patients With Cardiac Implantable Electronic Devices Undergoing Defibrillation Threshold Testing
Brief Title: Myocardial Injury in Patients With Cardiac Implantable Electronic Devices Undergoing Defibrillation Threshold Testing
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Allan S. Jaffe, Principal Investigator, Mayo Clinic
Other Study IDs: 19-008297
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2025-07-07 (Actual); Status verified 2025-07

CONDITIONS: ICD
Keywords: Defibrillation Threshold Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum or plasma samples remaining after initial analysis will be frozen and stored at -80 degrees Celsius for 120 months (10 years). These samples may be used if there are new and more sensitive biomarkers of myocardial injury that become available.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Researchers are trying to determine if heart injury occurs in patients with a cardiac implantable electronic device (CIED) who undergo a defibrillation threshold testing (DFT) procedure.

DETAILED DESCRIPTION:
CIED devices that deliver defibrillation can provide life-saving therapy to patients who have cardiac conditions that make them prone to develop a serious arrhythmia. Currently, there are two main CIED devices that deliver defibrillation therapy - transvenous internal cardioverter-defibrillator (ICD) and subcutaneous ICD. Conventional wisdom indicates that defibrillation causes myocardial injury. However, some studies including one by the present investigators have reported that external direct current cardioversion does not result in myocardial injury. There have been studies showing that ICD shocks results in myocardial injury. The concern with previous studies using transvenous ICDs is that the measurement of injury was done during DFT testing at the time of ICD implantation or when the patient came into hospital after an ICD shock. The confounder with DFT testing is that myocardial injury could have occurred during ICD implantation when the lead is screwed into the myocardium rather than during the testing. With hospitalization, the precipitating event that caused the arrhythmia stimulating the ICD discharge (e.g. an acute coronary syndrome) might also be the cause of myocardial injury. We plan to eliminate these confounders by recruiting patients who are undergoing a DFT procedure electively, remote from their ICD implantation date or clinical events.

In terms of the subcutaneous ICD implantation (in which the leads are not screwed into the myocardium), there is little data about myocardial injury when a shock is delivered. The investigators will attempt to determine if subcutaneous ICD shocks cause myocardial injury by assessing their troponin levels at the time DFT is performed during implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing elective defibrillation threshold testing of their transvenous ICD or defibrillation threshold testing of the subcutaneous ICD at the time of implantation

Exclusion Criteria:

* Patients under age 18
* Patients with myocardial infarction, coronary artery bypass grafting or any invasive cardiac procedure in the previous six weeks
* Pregnant patients
* Patients who cannot provide informed consent because of cognitive dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult males and females age 18 and above who have a cardiac implantable electronic device (CIED) or about to receive a CIED, and scheduled to undergo a defibrillation threshold testing (DFT).
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Myocardial injury | Baseline, approximately 6-24 hours after DFT procedure
  Changes in the high sensitivity cardiac troponin T (hs-cTnT) or troponin I (hs-cTnI) assay

CONTACTS AND LOCATIONS:
Overall Officials: Allan S Jaffe, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No